CLINICAL TRIAL: NCT02417298
Title: Ketamine Infusion for Acute Sickle Cell crisiS in the Emergency Department
Acronym: KISS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility
Sponsor: Billy Sin (Other)
Responsible Party: Sponsor-Investigator, Billy Sin, Primary investigator, The Brooklyn Hospital Center
Organization: The Brooklyn Hospital Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 668842
Record Dates: First submitted 2015-03-25; First posted 2015-04-15 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Pain; Sickle Cell Disorder
Keywords: ketamine; pain; sickle cell disorder
MeSH Terms: conditions — Pain; Anemia, Sickle Cell | interventions — Saline Solution; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Active Comparator): Ketamine 0.3 mg/kg intravenous push followed by ketamine infusion at 0.1 mg/kg/hr for 3 hours
  Interventions: Drug: Ketamine
- Saline (Placebo Comparator): Normal saline intravenous push (with volume to be administered equivalent to that of ketamine 0.3mg/kg, if the patient was to receive ketamine) followed by a normal saline infusion at the same rate as ketamine arm
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Normal saline — Normal saline intravenous push (with volume to be administered equivalent to that of ketamine 0.3mg/kg, if the patient was to receive ketamine) followed by a normal saline infusion at the same rate as ketamine arm
  Arms: Saline
Drug: Ketamine — 0.3mg/kg IVP ketamine followed by 0.1mg/kg/hr of ketamine infusion for 3 hours
  Arms: Ketamine

SUMMARY:
Pain associated with sickle cell disease is a common emergency department visit. It is also frequently associated with a high emergency department recidivism rate for pain control and admissions to the hospital. Opiates are considered the first line therapy for acute flares and to manage chronic pain. This often times leads to a stigma of being "opiate seekers" or "frequent fliers". With this study, we wish to explore whether adding ketamine to standard acute opiate therapy (morphine or dilaudid) will decrease subsequent repeat doses of opiates while improving the patient's perception of pain. In addition, we will be exploring whether ketamine as an adjuvant therapy can help reduce hospital admissions for the management of acute sickle cell crisis pain.

DETAILED DESCRIPTION:
The total number of required patients would be 53 per arm (106 patients). The targeted study population is patients who are 18 years old or older presenting with acute sickle cell crisis pain either described as diffuse throughout the body or localized to extremity/back. The expected duration of the study is 2 years

Prior to initiation of study, the research associates would be responsible for the randomization process. The goal of this study is to enroll 106 patients total (53 per arm). Patients will be assigned to a study arm via an online random-number generator (http://www.randomization.com). Each number will correlate to a sealed opaque envelope, which will be pulled in sequential order as patients are enrolled. Within each envelope will contain the particular study medication. A primary master list will be kept in a locked and secured cabinet in pharmacy. Only pharmacy personnel and the primary/secondary investigators will have access to this list. Pharmacy will use this master list to prepare study medications. A second master list would also be secured in the EM research room for back-up purposes. The secondary master list would be assessed only if the primary master list is lost. Only the primary and secondary investigator will have access to the secondary master list.

Detailed study procedures:

Step 1: Identification of patients with chief complaints or visit reasons of sickle cell via the Emergency Department's Statusboard by Research Associate or study investigators.

Step 2: Screening of potentially eligible patients with inclusion/exclusion criteria checklist as per Data Collection instrument (See attached Form 1) by Research Associate or study investigators.

Step 3: If patient is eligible, Research Associate or study investigators would obtain informed consent and explain potential risks and benefits with receiving study interventions.

Step 4: There will be no placebo only arm. All providers, except pharmacy, will be blinded to whether the patient is receiving ketamine or saline. All patients will receive conventional standard therapy (dilaudid or morphine) which will be ordered by the emergency department resident or attending. Each patient will receive an IVP bolus with infusion and a separate IVP. Arm A will include 0.3 mg/kg IVP bolus of Ketamine followed by a 0.1 mg/kg/hr infusion for 3 hours along with an initial dose of standard therapy. Arm B will receive a IVP bolus of normal saline (utilizing the 0.3 mg/kg calculation) followed by a normal saline infusion and then a separate standard therapy dose.

Step 5: An order would be placed by the medical resident, medical attending, a study investigator who is a physician, or a pharmacist under the permission of the attending physician into Allscripts for a study intervention.

Step 6: Upon receiving the order in Allscripts, the order would be verified by the pharmacy. Once notified of which envelope has been pulled pharmacy will prepare a ketamine IVP bolus and infusion or NS IVP bolus and infusion. Conventional therapy will be pulled from the general ED accudose stock by the ED RN. ED personnel will obtain the infusion preparation from pharmacy. It will be labeled for the patient, with study number, but without other identifying marks. When the study medication is picked up, pharmacy will open the sealed envelope to confirm which medication arm was prepared in order to internally verify the correct preparation.

Step 7: The nurse assigned to the patient would administer the intervention.

Step 8: A research associate or a study investigator would approach the patient to assess and record primary outcomes, secondary outcomes at designed time intervals. The data will be recorded on the data collection instrument. If additional medication is requested by the patient, the orders would be placed by the medical resident or attending who are assigned to the patient in the ED.

Step 9: All data retrieved from the paper data collection sheets will be transcribed into an encrypted and password protected electronic database by the research associate.

• All patient identifiers would be de-identified in the database. All participants would be assigned a study participant number.This database would be stored in the Emergency Department faculty or research room. Only the research associates or study investigators would have access to the electronic database. The paper data collection sheets would be stored in a stationary and locked cabinet in the Emergency Department for safe keeping. At the end of the study, these records will be maintained according to the hospital's record-retention policy.

Step 10: At the end of study enrollment, the data will be analyzed. Blinding will be removed for final data analysis and compilation.

Step 11: At the conclusion of the study, the final results and conclusions would be presented to the IRB. All data recorded from paper would be shredded and destroyed. All data recorded on electronic databases would be deleted.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old and older presenting with acute sickle cell crisis pain either described as diffuse throughout the body or localized to joint/extremity/back
* Describes pain to be greater than or equal to 2 on the NRS
* Consents to IV access
* Provides informed consent

Exclusion Criteria:

* Receiving IM therapy only
* Standard therapy plan is not morphine or dilaudid
* Previous enrollment in study
* Documented fever or subjectively reported fever
* Complaint of chest pain or shortness of breath or abdominal pain or headache
* Suspicion for acute chest crisis
* Patients with history or acute diagnosis of subarachnoid hemorrhage/increased intracranial pressure
* Severe hypertension(≥180/100)
* History of CAD or hypertension
* Presence of/suspected for traumatic head injury with or without loss of consciousness
* Presence of/suspected for myocardial ischemia
* Presence of/suspected for alcohol intoxication
* Hemodynamic instability
* History of psychiatric disorders,
* Known or suspected pregnancy or breastfeeding
* Allergy to ketamine
* Administration of opioids in previous 4 hours
* Patients with language barriers
* Ilicit drug use within the past 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11; Primary Completion 2018-04-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Change in patient's perception of pain | At baseline, 30, 60, 90, 120, 150 and 180 min after administration of intervention
  Pain will be assessed via the Numeric Rated Scale (NRS)
Total number of patients requiring hospital admission | 180 min after administration of intervention
  At the end of the study (180 minutes after initial administration of intervention) the number of patients requiring hospital admission will be quantified

SECONDARY OUTCOMES:
Change in patient perception of pain after discharge | 24 and 72 hours post ED discharge
  Pain will be assessed via the Numeric Rated Scale (NRS)
Total opiate consumed | 0, 30, 60, 90, 120, 150, and 180 minutes after administration of study intervention
  If opiates were ordered as part of standard therapy for patient, the total amount of opiates consumed would be quantified
Post test of disability and functional outcomes using the Sickle Cell Pain Burden Interview (SCPBI) | 180 minutes after initial study intervention
Incidence of hypertension | 0, 30, 60, 90, 120, 150, and 180 minutes after administration of study intervention
Incidence of dissociative effects (characterized by hallucination, disorientation, confusion, agitation, delirium, dreams) | 0, 30, 60, 90, 120, 150, and 180 minutes after administration of study intervention
Incidence of nausea | 0, 30, 60, 90, 120, 150, and 180 minutes after administration of study intervention
Incidence of vomiting | 0, 30, 60, 90, 120, 150, and 180 minutes after administration of study intervention
Incidence of dizziness | 0, 30, 60, 90, 120, 150, and 180 minutes after administration of study intervention
Incidence of headache | 0, 30, 60, 90, 120, 150, and 180 minutes after administration of study intervention
Time to patient discharge from the initiation of intervention | At the end of study period (180 minutes after initiation of study intervention)
Patient satisfaction of pain control | At the end of study period (180 minutes after initiation of study intervention)
  To be assessed via a Likert Scale

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hochberg, MD, Principal Investigator — The Brooklyn Hospital Center
Locations (1):
- The Brooklyn Hospital Center, Brooklyn, New York, United States

REFERENCES:
- [Background] Neri CM, Pestieau SR, Darbari DS. Low-dose ketamine as a potential adjuvant therapy for painful vaso-occlusive crises in sickle cell disease. Paediatr Anaesth. 2013 Aug;23(8):684-9. doi: 10.1111/pan.12172. Epub 2013 Apr 9. PMID 23565738
- [Background] Jennings CA, Bobb BT, Noreika DM, Coyne PJ. Oral ketamine for sickle cell crisis pain refractory to opioids. J Pain Palliat Care Pharmacother. 2013 Jun;27(2):150-4. doi: 10.3109/15360288.2013.788599. Epub 2013 May 21. PMID 23692261
- [Background] Tawfic QA, Faris AS, Kausalya R. The role of a low-dose ketamine-midazolam regimen in the management of severe painful crisis in patients with sickle cell disease. J Pain Symptom Manage. 2014 Feb;47(2):334-40. doi: 10.1016/j.jpainsymman.2013.03.012. Epub 2013 Jul 12. PMID 23856095
- [Background] Zempsky WT, Loiselle KA, Corsi JM, Hagstrom JN. Use of low-dose ketamine infusion for pediatric patients with sickle cell disease-related pain: a case series. Clin J Pain. 2010 Feb;26(2):163-7. doi: 10.1097/AJP.0b013e3181b511ab. PMID 20090444
- [Background] Meals CG, Mullican BD, Shaffer CM, Dangerfield PF, Ramirez RP. Ketamine infusion for sickle cell crisis pain in an adult. J Pain Symptom Manage. 2011 Sep;42(3):e7-9. doi: 10.1016/j.jpainsymman.2011.06.003. No abstract available. PMID 21854993
- [Background] Uprety D, Baber A, Foy M. Ketamine infusion for sickle cell pain crisis refractory to opioids: a case report and review of literature. Ann Hematol. 2014 May;93(5):769-71. doi: 10.1007/s00277-013-1954-3. Epub 2013 Nov 15. PMID 24232306
- [Background] Yawn BP, Buchanan GR, Afenyi-Annan AN, Ballas SK, Hassell KL, James AH, Jordan L, Lanzkron SM, Lottenberg R, Savage WJ, Tanabe PJ, Ware RE, Murad MH, Goldsmith JC, Ortiz E, Fulwood R, Horton A, John-Sowah J. Management of sickle cell disease: summary of the 2014 evidence-based report by expert panel members. JAMA. 2014 Sep 10;312(10):1033-48. doi: 10.1001/jama.2014.10517. PMID 25203083